CLINICAL TRIAL: NCT03566147
Title: Treatment of Retinitis Pigmentosa and Leber Congenital Amaurosis by Primary Retinal Pigment Epithelial Cells Transplantation
Brief Title: Treatment of RP and LCA by Primary RPE Transplantation
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eyecure Therapeutics Inc. (Industry)
Collaborators: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TR-RPE-RP/LCA
Record Dates: First submitted 2018-06-12; First posted 2018-06-21 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-06

CONDITIONS: Leber Congenital Amaurosis, Retinitis Pigmentosa
MeSH Terms: conditions — Leber Congenital Amaurosis; Retinitis Pigmentosa | interventions — Cell Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low dose group (Experimental): 300,000 HuRPE cells
  Interventions: Biological: Human primary Retinal Pigment Epithelial (HuRPE) cells
- middle dose group (Experimental): 500,000 HuRPE cells
  Interventions: Biological: Human primary Retinal Pigment Epithelial (HuRPE) cells
- high dose group (Experimental): 1,000,000 HuRPE cells
  Interventions: Biological: Human primary Retinal Pigment Epithelial (HuRPE) cells

INTERVENTIONS:
Biological: Human primary Retinal Pigment Epithelial (HuRPE) cells — HuRPE will be transplanted by a board-certified vitreoretinal surgeon, which will be administered into the subretinal space of experimental eye through a standard surgical approach.

SUMMARY:
Early Phase I Study of the Safety and Preliminary Efficacy of Human primary Retinal Pigment Epithelial (HuRPE) Cells Subretinal Transplantation in Retinitis Pigmentosa (RP) and Leber Congenital Amaurosis (LCA) Patients

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of RP or LCA;
2. Experimental eye with best-corrected visual acuity (BCVA) of no more than 35 letters or visual field of less than 10 degree;
3. Patient understand and sign the consent form.

Exclusion Criteria:

1. Blood routine examination is abnormal (hemoglobin<10gm/dL; blood platelet count<100k/mm³; neutrophil count<1000/mm³)
2. Blood biochemistry is abnormal (ALT／AST>1.5; creatinine>1.3mg/dL)
3. Experimental eye has optic nerve atrophy caused by glaucoma
4. Experimental eye has retinal detachment, or has received retinal detachment surgery.
5. Patients with uveitis and other endophthalmitis
6. Patients with other ocular disease affecting vision.
7. Patients have participated in clinical study of ocular or systemic drug use in recent 6 months.
8. Patients with medical history of malignant cancer (except resected basal cell carcinoma and squamous-cell carcinoma).
9. Patients with medical history of myocardial infarction
10. Patient with diabetes
11. Patient with Parkinson disease or Alzheimer's disease
12. Patients are under the treatment of immunosuppressive agent (except intermittent, low-dose corticosteroid treatment).
13. Patients with other medical conditions that restricts the compliance and safety of patients, or affects experimental results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
best-corrected visual acuity (BCVA) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ningli Wang, Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No